CLINICAL TRIAL: NCT05875337
Title: The Effect of Acupressure on Procedural Pain, Anxiety and Hemodynamic Variables During Chest Tube Removal in Patients With Open Heart Surgery: A Double-Blind Randomized Controlled Trial
Brief Title: The Effect of Acupressure on Procedural Pain, Anxiety and Hemodynamic Variables During Chest Tube Removal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Tugba CAM YANIK, Research Assistant, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: MersinU.
Record Dates: First submitted 2023-05-15; First posted 2023-05-25 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Pain, Postoperative; Anxiety; Hemodynamic Instability
MeSH Terms: conditions — Pain, Postoperative; Anxiety Disorders | interventions — Acupressure

STUDY DESIGN:
Intervention Model Description: Double-blind randomized controlled experimental trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: In the study, a researcher (F.E.Ö.) will determine the acupressure and placebo points to be applied to the patients. However, the certified researcher (T.Ç.Y.) who will perform the acupressure and placebo application will perform the application without knowing whether these points are acupressure or placebo points and will be blinded. The participants will not know whether they are in the acupressure or placebo acupressure group. Thus, the research will be carried out as a double-blind randomized controlled trial. When the research is completed, the data of the acupressure and placebo acupressure groups (coded as A or B) will be transferred to the computer environment by a researcher independent of the research, and the data will be analyzed and reported by a statistician using blinded technique.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupressure Group (experimental) (Experimental): In the acupressure groups the points are LI4, LI11 and HT7.
  Interventions: Other: Acupressure
- Placebo Acupressure Group (control) (Placebo Comparator): In the placebo acupressure group the points are 1.5 cm away from LI4, LI11 and HT7 points.
  Interventions: Other: Placebo acupressure

INTERVENTIONS:
Other: Acupressure — Before starting the acupressure point application, the area around the area where the pressure will be applied for 20-30 seconds will be gently rubbed with the palm of the hand. By gently rubbing the surrounding tissue, tension and tissue sensitivity will be reduced and the tissue will be relaxed by heating, relaxing and preparing the point area. Pressure will be applied to the determined points (LI4, LI11 and HT7) with the thumb, index or middle finger manually for 5 seconds to create a depth of 1-1.5 cm and rest for 2 seconds. Each point will be applied for 2 minutes and the application will last 12 minutes.
  Arms: Acupressure Group (experimental)
Other: Placebo acupressure — Before starting the application to the placebo acupressure point, the area around the area where pressure will be applied for 20-30 seconds will be gently rubbed with the palm of the hand. By gently rubbing the surrounding tissue, tension and tissue sensitivity will be reduced and the tissue will be relaxed by heating, relaxing and preparing the point area. Light pressure will be applied to the determined points (1.5 cm away from LI4, LI11 and HT7 points) with the thumb, index or middle finger. Each point will be applied for 2 minutes and the application will last 12 minutes.
  Arms: Placebo Acupressure Group (control)

SUMMARY:
When the literature was reviewed, many studies were found in which various non-pharmacologic interventions such as reflexology, music therapy, slow and deep breathing exercises, relaxation exercises and cold application were examined in the control of pain associated with chest tube removal. However, a limited number of studies have examined the effect of acupressure on the control of pain caused by chest tube removal; there are no studies in which LI4, LI11 and HT7 acupressure points were used and anxiety level and hemodynamic variables were examined along with procedural pain. Thus, the aim of this study was to investigate the effect of acupressure on procedural pain, anxiety and hemodynamic variables after chest tube removal after open heart surgery.

DETAILED DESCRIPTION:
Before starting the acupressure/placebo acupressure point application, the area around the area where pressure will be applied for 20-30 seconds will be gently rubbed with the palm of the hand. By gently rubbing the surrounding tissue, tension and tissue sensitivity will be reduced and the tissue will be relaxed by heating, relaxing and preparing the point area. Pressure will be applied to the determined points (LI4, LI11 and HT7 or points 1.5 cm away) with the thumb, index or middle finger manually for 5 seconds to create a depth of 1-1.5 cm, and rest for 2 seconds. Each point will be applied for 2 minutes and the application will last 12 minutes.

When acupressure/plesebo acupressure application is completed, the chest tube will be removed by the physician. Procedural pain level, anxiety level and hemodynamic variables of all patients in the acupressure and placebo acupressure groups will be re-evaluated immediately and 15 minutes after removal of the chest tube.

ELIGIBILITY:
Inclusion Criteria:

* With only one chest tube after open heart surgery,
* 18 years of age or older,
* Conscious and cooperative,
* Speaks and understands Turkish,
* General condition and hemodynamic variables are stable,
* Planned surgical intervention,
* No previous chest tube experience,
* Acupressure/placebo acupressure without scars, scars, tenderness in the area to be acupressure,
* No active COVID-19 infection,
* Does not have any psychiatric diagnosis,
* Not using psychiatric and/or local neuromuscular blocking drugs,
* Patients who agreed to participate in the study (signed the Informed Consent Form)

Exclusion Criteria:

* No chest tube or multiple chest tubes after open heart surgery,
* Under 18 years of age,
* Conscious and uncooperative,
* Speaking Turkish but not understanding it,
* Unstable general condition and hemodynamic variables,
* Underwent emergency surgical intervention,
* Anyone with previous chest tube experience,
* Wounds, scars, tenderness in the area where acupressure/placebo acupressure will be applied,
* With active COVID-19 infection,
* Has an existing psychiatric diagnosis,
* Psychiatric and/or local neuromuscular blocking drugs,
* Patients who did not agree to participate in the study (did not sign the Informed Consent Form).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2023-05-25 (Actual); Primary Completion 2023-05-25 (Actual); Study Completion 2024-05-25 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Pain on the Visual Analog Scale at 15 minutes | Baseline and 15 minutes
  The VAS, which is a safe, easily applicable scale tool generally accepted in the literature, consists of a 10 cm long line and subjective descriptive statements at both ends of the scale (0 cm=none and 10 cm=highest degree of presence). The individual marks the appropriate place on the scale on this 10 cm line. The distance from the beginning of the scale to the mark is measured with a ruler and the pain level of the individual is determined numerically in cm.

SECONDARY OUTCOMES:
Change from baseline in Anxiety on the State Anxiety Inventory at 15 minutes | Baseline and 15 minutes
  The total score of the scale is calculated by subtracting the total weighted score of the inverted statements from the total weighted score of the direct statements and adding the number 50, which is the predetermined and unchanging value of the State Anxiety Inventory. A score of 30 and above on this scale indicates moderate anxiety and a score of 45 and above indicates severe anxiety.
Change from baseline in SpO2 at 15 minutes. | Baseline and 15 minutes.
  Oxygen saturation measured at the specified times will be recorded for the acupressure and placebo acupressure group patients. Hemodynamic variables will be monitored and recorded with a bedside monitor (Nihon Kohden, Tokyo). To ensure data reliability and accuracy, these monitors are calibrated monthly by the biomedical engineering department as per hospital policy.
Change from in respiration rate at 15 minutes. | Baseline and 15 minutes
  Respiration rate measured at the specified times will be recorded for the acupressure and placebo acupressure group patients. Hemodynamic variables will be monitored and recorded with a bedside monitor (Nihon Kohden, Tokyo). To ensure data reliability and accuracy, these monitors are calibrated monthly by the biomedical engineering department as per hospital policy.
Change from in systolic blood pressure at 15 minutes | Baseline and 15 minutes
  Systolic blood pressure measured at the specified times will be recorded for the acupressure and placebo acupressure group patients. Hemodynamic variables will be monitored and recorded with a bedside monitor (Nihon Kohden, Tokyo). To ensure data reliability and accuracy, these monitors are calibrated monthly by the biomedical engineering department as per hospital policy.
Change from in diastolic blood pressure at 15 minutes. | Baseline and 15 minutes
  Diastolic blood pressure measured at the specified times will be recorded for the acupressure and placebo acupressure group patients. Hemodynamic variables will be monitored and recorded with a bedside monitor (Nihon Kohden, Tokyo). To ensure data reliability and accuracy, these monitors are calibrated monthly by the biomedical engineering department as per hospital policy.
Change from in heart rate at 15 minutes. | Baseline and 15 minutes
  Heart rate measured at the specified times will be recorded for the acupressure and placebo acupressure group patients. Hemodynamic variables will be monitored and recorded with a bedside monitor (Nihon Kohden, Tokyo). To ensure data reliability and accuracy, these monitors are calibrated monthly by the biomedical engineering department as per hospital policy.

CONTACTS AND LOCATIONS:
Overall Officials: Gülay ALTUN UĞRAŞ, PhD, Study Director — Mersin University; Serpil YÜKSEL, PhD, Principal Investigator — Necmettin Erbakan University; Didem KANDEMİR, PhD, Principal Investigator — England
Locations (1):
- Mersin University Hospital, Mersin, Yenişehir, Turkey (Türkiye)